CLINICAL TRIAL: NCT00500981
Title: Do Internal Jugular Vein Measurements Made By Ultrasound Correlate With Fluid Responsiveness in Ventilated Post-Operative Cardiac Surgical Patients?
Brief Title: Internal Jugular Vein Ultrasound Measures and Fluid Responsiveness in Post-Operative Cardiac Surgical Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Department of Critical Care Medicine (Unknown)
Responsible Party: Principal Investigator, Dr. Dan Zuege, Clinical Associate Professor of Medicine, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20855
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Fluid Therapy; Cardiac Surgical Procedures
Keywords: Fluid responsiveness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous fluid bolus (Experimental): Administration of 500 ml of 10% pentastarch
  Interventions: Procedure: Volume challenge; Procedure: Ultrasound evaluation of internal jugular vein

INTERVENTIONS:
Procedure: Volume challenge
Procedure: Ultrasound evaluation of internal jugular vein

SUMMARY:
The goal of this study is to evaluate whether measures of the size of the internal jugular vein have clinical utility in predicting whether patients may benefit from treatment with intravenous fluid.

DETAILED DESCRIPTION:
The optimal therapy for numerous disease states involves the replenishment of intravascular volume. Unfortunately, our current clinical measures of volume status are imperfect. Given biologic plausibility and preliminary study, it is possible that static and/or dynamic measures of internal jugular vein (IJV) size may correlate with volume status and/or be associated with volume responsiveness. If so, this type of assessment might be a more ideal clinical volume-assessment tool. This pilot study aims to establish proof of concept via evaluation of this question in patients following cardiac surgery.

This is a prospective observational study of physiologically-stable, ventilated patients post-cardiac surgery. The primary objective of this study is to evaluate the relationship between the static size of the right IJV and fluid responsiveness in ventilated post-operative cardiac surgical patients. A secondary objective is to evaluate the relationship between dynamic variations in the size of the right IJV related to respiration and leg-raising and fluid responsiveness in the same group. Static and dynamic ultrasound measurements of the right IJV will be performed pre-volume challenge.

Volume responsiveness will be independently assessed by cardiac index measurement before and after rapid infusion of 10% pentastarch. 30 subjects will be recruited pre-operatively and informed consent obtained. Stability of sedation, mechanical ventilation, and hemodynamics will be assured prior to initiation of measurements. Baseline static and respiratory dynamic ultrasound measurements of the right IJV will be obtained and then repeated after bilateral leg-raising. Baseline hemodynamics and cardiac outputs will be obtained using indwelling pulmonary artery catheters. A standardized volume challenge of 10% pentastarch given over 15 minutes will then be provided followed by repeat hemodynamic and cardiac output measurements.

Offline measurements of IJV size will be obtained from unmodified stored video loops by a single observer blinded to patient identity, hemodynamic, and fluid response data. Fluid responsiveness will be assessed by examining the change in cardiac index after volume challenge with a fluid responsive state defined as an increase of ≥ 12 % of cardiac index after volume challenge. The relationship between volume responsiveness and IJ ultrasound measures will be evaluated continuously and dichotomously.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old)
* Able to provide advanced informed consent
* Planned elective or semi-urgent cardiac surgery

Exclusion Criteria:

* Severe tricuspid regurgitation or planned tricuspid valve surgery
* Congenital heart disease associated with cardiac shunting
* Pre or post-operative presence of an intra-aortic balloon pump
* Severe chronic obstructive pulmonary disease
* Hemodynamic instability such that inotropes/vasopressor dosing is not constant
* Respiratory instability and/or need for PEEP > 5 cmH20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between the static size of the right IJV and fluid responsiveness in ventilated post-operative cardiac surgical patients. | 1 hour

SECONDARY OUTCOMES:
To evaluate the relationship between dynamic variations in the size of the right IJV related to respiration and leg-raising and fluid responsiveness in ventilated post-operative cardiac surgical patients. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zuege, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada